CLINICAL TRIAL: NCT02228811
Title: A Multicenter Phase 1 Ascending Dose Study of DCC-2701 To Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Patients With Advanced Solid Tumors
Brief Title: A Study of DCC-2701 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2701-01-001
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2016-12

CONDITIONS: Locally Advanced Tumors; Metastatic Solid Tumors; Cancers With MET Genomic Alterations; Cancers With TRK Genomic Alterations
MeSH Terms: interventions — DCC-2701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCC-2701 tablet (Experimental): DCC-2701 tablets in escalating dose cohorts given orally BID (twice daily) every 12 hours for a 28-day cycle. Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: DCC-2701 tablet

INTERVENTIONS:
Drug: DCC-2701 tablet

SUMMARY:
The main purpose of this study is to investigate the safety of the investigational drug DCC-2701 and whether it will work to help people who have advanced solid tumors or cancer that has spread to other parts of the body.

DETAILED DESCRIPTION:
This is a first-in-human study of DCC-2701. The primary purpose of this study is to determine what dose of DCC-2701, can be given safely to patients with advanced solid tumors.

The study will have two phases. The first phase will assess escalating doses of DCC-2701 in order to determine the maximally tolerated dose (MTD) and the optimal dosing regimen (ODR) of DCC-2701. Once the MTD and ODR is established, a dose expansion phase will further evaluate the safety of DCC-2701, as well as the activity of DCC-2701 in select solid tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumor that has progressed or was not responsive to standard therapy
* The cancer has no proven effective therapy
* The cancer can be biopsied (depending on the tumor type and/or the dose of drug received, tumor biopsies may be required)
* Able to swallow tablets

Exclusion Criteria:

* Have active central nervous system (CNS) metastasis
* Have an active infection of any kind (fungal, viral, or bacterial)
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of DCC-2701 | 28 days (1 cycle)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of DCC-2701 | Cycle 1: Predose and up to 24 hours postdose (Cycle = 28 Days)
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of DCC-2701 | Cycle 1: Predose and up to 24 hours postdose (Cycle = 28 Days)
Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of DCC-2701 | Cycle 1: Predose and up to 24 hours postdose (Cycle = 28 Days)
Number of Participants with Tumor Response according to Response Evaluations Criteria in Solid Tumors (RECIST) version 1.1 | Baseline through study completion (estimated as 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Rosen, M.D., Study Director — Deciphera Pharmaceuticals, LLC
Locations (5):
- United States (5):
  - University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas